CLINICAL TRIAL: NCT06307067
Title: Improving Care for Uncomplicated URinary Tract Infection-associated Symptoms in Primary Healthcare Settings in INDOnesia
Acronym: URINDO
Status: Not yet recruiting | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Saiful Anwar Hospital (Other); Brawijaya University, Malang, Indonesia (Unknown); Diponegoro University/Diponegoro National Hospital, Semarang, Indonesia (Unknown); Bali Mandara Hospital, Denpasar, Bali, Indonesia (Unknown)
Responsible Party: Principal Investigator, Juliëtte Severin, Associate professor, Medical coordinator Unit infection prevention, Erasmus Medical Center
Other Study IDs: URINDO
Record Dates: First submitted 2024-03-06; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Urinary Tract Infections
Keywords: antimicrobial use; diagnostic test
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — Bacteria from urine culture
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-intervention group: patients being treated according to the old method (no dipstick as diagnostic test)
- Post-intervention group: patients being treated according to the new method (dipstick as diagnostic test)
  Interventions: Diagnostic Test: Urine dipstick

INTERVENTIONS:
Diagnostic Test: Urine dipstick — Urine dipstick is a point of care test that can be performed on the urine in the public health center.
  Groups: Post-intervention group

SUMMARY:
In the present study, we aim to analyze the impact of the introduction of a urinary dipstick test for patients presenting with uncomplicated UTI-associated symptoms on antibiotic prescription in primary health care in Indonesia. In addition, the knowledge of HCW regarding antibiotics and prudent use of antibiotics in the community setting will be investigated.

Specific aims of the study:

1. To analyze the quality of antibiotic prescriptions for uncomplicated UTI in the primary health care settings in Indonesia, before introduction of urinary dipstick testing compared to after introduction of urinary dipstick testing.
2. To analyze the knowledge level of healthcare workers on uncomplicated UTI and prudent antibiotic use in primary health care settings in Indonesia.

DETAILED DESCRIPTION:
Uncomplicated urinary tract infection (UTI) is one of the most frequent diagnoses and reasons for prescribing antibiotics in primary health care, however the laboratory capacity to perform urine cultures in primary health care in Indonesia is limited. Consequently, inappropriate antibiotic prescriptions for uncomplicated UTI patients in the primary health care may occur.

A before-after study will be carried out in primary health care settings in three cities (Malang, Semarang, and Denpasar) in Indonesia.

The specific aims will be addressed as follows:

Aim 1:

The study will be divided into three phases: pre-intervention (3 months) (i.e. in which patients are being treated according to the old method), intervention (1 month) (i.e., wash-in period, HCW will be trained to conduct the urinary dipstick test), and post-intervention (3 months) (i.e. in which for all patients with urinary complaints a dipstick test will be used). Urinary dipstick testing will be introduced as an intervention to rule-out uncomplicated UTI in the primary health care. Urine culture will be performed to confirm the diagnosis of uncomplicated UTI based on the bacterial colony count on the MacConkey agar. Urine specimen will be inoculated on to MacConkey agar and stored in 2-8oC until incubating in the microbiology laboratory of Dr. Saiful Anwar hospital (Malang), Diponegoro National hospital (Semarang), or Bali Mandara hospital (Denpasar). Identification of isolates and antimicrobial susceptibility testing will be performed using Vitek2 (bioMérieux). The urine culture results will not change the decision of antibiotic therapy to the patients.

Qualitative evaluation of antibiotics for uncomplicated UTI in primary health care settings will be performed by the Gyssens' algorithm and subsequent comparison before (pre-intervention) and after urinary dipstick testing (post-intervention) was applied (Hadi U, et al, 2008). All adult patients with uncomplicated UTI are eligible for inclusion in the study. Of each included patient, we will collect the following information after written consent: basic characteristics (e.g., gender, age) and UTI complaints (e.g. dysuria and lower abdominal pain) by structured interview. Participants will provide a clean-catch mid-stream urine for (dipstick test and) culture. However, patients who have recurrent episodes of uncomplicated UTI, pregnant women, and patients with recent antibiotic use (any antibiotic use within 3 months before visit) will be excluded. We will ask patients to return to the same public health center within one week after inclusion if they have the same complains, this will be recorded.

Sample size: 50 patients in each group; this would lead to a total sample size of 300 patients.

Aim 2:

The knowledge on and current practice of uncomplicated UTI management in primary health care settings will be obtained by a survey among HCW in the baseline phase (pre-intervention). The survey will be partly open-ended questions including the number of uncomplicated UTI cases per month (on average), the complaints of patient with uncomplicated UTI, how the healthcare workers decide to treat and not to treat for patients with suspected uncomplicated UTI, what antibiotics the healthcare workers choose and why they choose that kind of antibiotics. General knowledge on antibiotics will also be measured.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients with uncomplicated urinary tract infection

Exclusion Criteria:

patients who have recurrent episodes of uncomplicated UTI, pregnant women, and patients with recent antibiotic use (any antibiotic use within 3 months before visit)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female and male patients will be included, but women suffer more from uncomplicated UTI.
Study Population: Patients that come to a public health center with symptoms of an uncomplicated urinary tract infection
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-11-04 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
appropriateness of prescriptions for uncomplicated UTI-associated symptoms in the primary health care settings in Indonesia | 2024

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided